CLINICAL TRIAL: NCT04453280
Title: Antibody Detection in COVID-19 Cured Patients (SARS-CoV-2-CZ-Immunity)
Acronym: SARSCoV2CZImun
Status: Completed | Type: Observational
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: Ministry of Health, Czech Republic (Other Government); Masaryk University (Other); Institute for Clinical and Experimental Medicine (Other Government); Brno University Hospital (Other); St. Anne's University Hospital Brno, Czech Republic (Other); Masaryk Memorial Cancer Institute (Other); Regional Public Health Office of the South Moravian Region based in Brno, Czech Republic (Unknown); Public Health Office of the Capital City of Prague, Czech Republic (Unknown); Regional Public Health Office of the Central Bohemian Region based in Prague, Czech Republic (Unknown)
Responsible Party: Sponsor
Other Study IDs: UZIS 2020/2
Record Dates: First submitted 2020-06-30; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: COVID; SARS-CoV-2
Keywords: SARS-CoV-2; antibody; humoral immunity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma sampling will be archived in the biobank for subsequent quantitative analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 - Prague and Central Bohemian Region: A population cohort of cured patients based on epidemiologically defined demographic parameters - Prague and Central Bohemian Region population
  Interventions: Diagnostic Test: Quantitative analysis of anti-SARS-CoV-2-antibodies; Diagnostic Test: SARS-CoV-2 diagnostic rapid test
- Cohort 2 - South Moravian Region: A population cohort of cured patients based on epidemiologically defined demographic parameters - South Moravian Region population.
  Interventions: Diagnostic Test: Quantitative analysis of anti-SARS-CoV-2-antibodies

INTERVENTIONS:
Diagnostic Test: Quantitative analysis of anti-SARS-CoV-2-antibodies — Plasma sampling will be collected and archived for subsequent quantitative analysis of anti-SARS-CoV-2 antibodies - IgG, IgM and IgA.
Diagnostic Test: SARS-CoV-2 diagnostic rapid test — The rapid test detects the presence of antibodies against SARS-CoV-2 by the immunochromatographic reaction.
  Groups: Cohort 1 - Prague and Central Bohemian Region

SUMMARY:
The aim of the SARS-CoV-2-CZ-Immunity study is to determine the time profile of the presence of antibodies against SARS-CoV-2 in blood plasma by quantification of antibodies or performing a rapid test in COVID-19 cured patients.

DETAILED DESCRIPTION:
COVID-19 is caused by a new type of coronavirus called SARS-CoV-2. It is a highly infectious disease, manifested mainly by fever, respiratory problems, muscle pain, and fatigue. However, despite the publication of hundreds of papers in the literature, fundamental information about the spread and course of the disease is still lacking in COVID-19. One of such key information is the time profile of the presence of antibodies against SARS-CoV-2 after the disease.

The SARS-CoV-2-CZ-Immunity study is aiming at the determination of the time profile of the presence of antibodies against SARS-CoV-2 in blood plasma by quantification of antibodies or performing a rapid test in COVID-19 cured patients.

ELIGIBILITY:
Inclusion Criteria:

* signed Informed Consent
* residing in Prague, Central Bohemian Region or South Moravian Region
* demographic criteria: persons aged 8-17 and persons aged 18 and more
* clinical criteria: (i) diagnosis of COVID-19 confirmed by PCR (ii) cured patients: clearance of SARS-CoV-2 viral RNA demonstrated by two consecutive negative RT-PCR results (iii) without acute health problems

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Both cohorts will be selected from all actually cured individuals from specific demographic areas described in the cohorts. The cohorts of people will be addressed by Public Health Office.
Sampling Method: Non-Probability Sample
Enrollment: 695 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2020-06-03 (Actual); Study Completion 2020-06-03 (Actual)

PRIMARY OUTCOMES:
Determination of the concentration of anti-SARS-CoV-2 antibodies in relation to the categories of cured patients. | May 2020
  The primary outcome is the determination of the concentration of anti-SARS-CoV-2 antibodies IgG, IgM, and IgA classes in relation to the categories of cured patients according to the time from the date of cure from the COVID-19 disease to the date of examination.

SECONDARY OUTCOMES:
Determination of the concentration of anti-SARS-CoV-2 antibodies in relation to the age and to the severity of the disease. | June 2020
  The determination of the concentration of anti-SARS-CoV-2 antibodies IgG, IgM, and IgA classes in relation to the categories of cured patients according to their age: category 8-17, 18-39, 40-59, 60 and more years and according to the severity of the disease.
The quantification of the dependence of the change in the concentration of anti-SARS-CoV-2 antibodies. | June 2020
  The quantification of the dependence of the change in the concentration of anti-SARS-CoV-2 antibodies IgG, IgM, and IgA classes on the time since cure (analysis by statistical model)

OTHER OUTCOMES:
The identification of potential donors of convalescent plasma. | June2020
  The identification of individuals in the study population, who can be contacted as voluntary donors of convalescent plasma, which is one of the therapeutic modalities in patients with severe COVID-19 disease.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Prymula, Prof., Principal Investigator — Ministry of Health, Czech Republic; Jarmila Rážová, M.D., Ph.D., Principal Investigator — Ministry of Health, Czech Republic; Ladislav Dušek, Prof., Principal Investigator — Institute of Health Information and Statistics of the Czech Republic; Dalibor Valík, Prof., Principal Investigator — Masaryk Memorial Cancer Institute
Locations (1):
- Institute of Health Information and Statistics of the Czech Republic, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.